CLINICAL TRIAL: NCT03566693
Title: Continuous Glucose Monitoring (CGM) in Type 2 Diabetes (T2D) Basal Insulin Users: The Mobile Study (MOBILE)
Brief Title: Type 2 Diabetes (T2D) Basal Insulin Users: The Mobile Study (MOBILE)
Acronym: MOBILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DexCom, Inc. (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTL-902822
Record Dates: First submitted 2018-06-01; First posted 2018-06-25 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continous Glucose Monitor (Experimental)
  Interventions: Device: Dexcom G6 CGM System
- Self Monitoring Blood Glucose (Active Comparator)
  Interventions: Device: Blood glucose meter

INTERVENTIONS:
Device: Dexcom G6 CGM System — continuous glucose monitor
  Arms: Continous Glucose Monitor
Device: Blood glucose meter — Blue-tooth enabled blood glucose meter
  Arms: Self Monitoring Blood Glucose

SUMMARY:
A study to compare the glycemic and quality of life benefits of diabetes management using Dexcom G6 continuous glucose monitoring (CGM) or self-monitored blood glucose (SMBG) made by study participants and their primary care physicians. Decisions will be based on insights from real-time use and retrospective insights, determined during remote visits.

Participants will have type 2 diabetes and be using basal insulin (with or without oral medications and/or Glucagon-Like-Peptide-1 (GLP-1) analogue) and have an elevated Hemoglobin A1C (HbA1c).

DETAILED DESCRIPTION:
The study is referred to as the "Continuous Glucose MOnitoring in T2D Basal InsuLin UsErs, also known as The MOBILE Study" and will assess potential benefits of using Continuous Glucose Monitoring (CGM) versus traditional Blood Glucose Monitoring (BGM) in people with Type 2 Diabetes using basal insulin with or without oral medications and who have an elevated HbA1c between 7.8 -11.5%. In this study, the investigator's role is largely advisory, providing insights and interpretations of the glucose data obtained from BGM or CGM devices and formally communicating medication recommendations to the participant and their treating community clinician. Participants will be recruited from outside of the investigator team's diabetes and endocrine practice.

The protocol comprises of 2 studies: the 1st study (also called Phase 1) will evaluate the values of CGM after eight months of use. The 2nd study (also called Phase 2) will evaluate if any glycemic benefits attained in study one are sustainable for an additional six months.

At the time of enrollment, participants will undergo a run-in period of blinded CGM for a duration of 10 days. Baseline Patient Report Outcome (PRO) tools and surveys will be administered at time of enrollment.

The study design includes two phases. During Phase 1, participants with T2D taking basal insulin will be randomized into two groups - CGM Group or SMBG Group. Phase 1 is of 8 months duration. The CGM group will comprise of 4 scheduled clinic visits: at week 2, month 1, month 3, and month 8. The SMBG group will comprise of 5 scheduled clinic visits: at week 2, month 1, month 3, pre-month 8 and month 8. Both groups will have structured phone/remote visits at months 2, 4 and 6 during which glucose data will be reviewed and summarized. HbA1c will be measured at baseline, 3 months and 8 months. Participants will complete PRO tools and surveys at 8 months.

Phase 2 will consist of 3 groups: participants continuing use of SMBG since the beginning of Phase 1; participants re-randomized from the Phase 1 CGM Group and assigned to SMBG; participants re-randomized from Phase 1 CGM Group and assigned to CGM. Phase 2 duration is 6 months. This phase involves 1 phone contact and either 2 visits at Month 14 for SMBG participants to wear blinded CGM or one visit for CGM participants. HbA1c will be measured at 14 months. Participants will complete PRO tools and surveys at month 14. For all participants, study participation will end upon completion of month 14 visit .

ELIGIBILITY:
Major Inclusion Criteria:

* Age 30 or older
* Diagnosis of Type 2 diabetes
* HbA1c between 7.8-11.5%
* Use of basal insulin, with or without concomitant use of oral agents or GLP-1 agonist

Major Exclusion Criteria:

* Pregnancy
* Renal disease
* Conditions that impact the stability of a HbA1c measurement
* Use of prandial insulin

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Phase 1: Change in HbA1c | Baseline to Month 8
  Phase 1: Between group differences (CGM and SMBG) for the change in HbA1c (from Central Lab) from baseline to Month 8
Phase 2: Change in CGM time in target range | Month 8 to Month 14
  Between group differences for the Phase 1 CGM Group re-randomized to Discontinue CGM (use SMBG only) or to Continue CGM for the change in time in target range (70-180 mg/dL) from Month 8 to Month 14

SECONDARY OUTCOMES:
Phase 1: Change in CGM time in target range | Baseline to Month 8
  Between group differences (CGM and SMBG) from baseline to Month 8 of change in CGM time in target range 70-180 mg/dL
Phase 1: Change in CGM time-hyperglycemic | Baseline to Month 8
  Between group differences (CGM and SMBG) from baseline to Month 8 of change in CGM time-hyperglycemic, defined as >250 mg/dL
Phase 1: Change in mean glucose from CGM | Baseline to Month 8
  Between group differences (CGM and SMBG) from baseline to Month 8 of change in mean glucose from CGM
Phase 1: Percent decreasing HbA1c by ≥0.5% | Baseline to Month 8
  Between group differences (CGM and SMBG) from baseline to Month 8 of percent decreasing HbA1c by ≥0.5% (absolute)
Phase 1: Proportion increasing CGM time in target range by ≥10% and ≥15% | Baseline to Month 8
  Between group differences (CGM and SMBG) from baseline to Month 8 of proportion increasing CGM time in target range by ≥10% and ≥15% (absolute)
Phase 1: Percent adding or removing diabetes medications | Baseline to Month 8
  Between group differences (CGM and SMBG) from baseline to Month 8 of percent adding or removing diabetes medications (starting or stopping medications)
Phase 1: Change in HbA1c based on their baseline HbA1c | Baseline to Month 8
  Between group differences (CGM and SMBG) from baseline to Month 8 of change in HbA1c based on their baseline HbA1c (restricted to participants with baseline HbA1c ≥8.5%,≥9.0%, ≥9.5%, ≥10.0%)
Phase 1: Change in CGM glucose variability | Baseline to Month 8
  Between group differences (CGM and SMBG) from baseline to Month 8 of change in CGM glucose variability measured by the coefficient of variation
Phase 1: Change in CGM time-hypoglycemic | Baseline to Month 8
  Between group differences (CGM and SMBG) from baseline to Month 8 of change in CGM time-hypoglycemic, defined as <70mg/dL
Phase 2: Change in HbA1c | Month 8 to Month 14 & Baseline to Month 14
  Between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM group from Month 8 to Month 14 and between group differences for the Continue CGM and the Continue SMBG groups from baseline to Month 14 of change in HbA1c (central lab)
Phase 2: Change in CGM time-hyperglycemic | Month 8 to Month 14 & Baseline to Month 14
  Between group differences (CGM and SMBG) from baseline to Month 8 of change in CGM time-hyperglycemic, defined as >250 mg/dL
Phase 2: Percent decreasing HbA1c by ≥0.5% | Month 8 to Month 14 & Baseline to Month 14
  Between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM group from Month 8 to Month 14 and between group differences for the Continue CGM and the Continue SMBG groups from baseline to Month 14 of percent decreasing HbA1c by ≥0.5% (absolute)
Phase 2: Proportion increasing CGM time in target range by ≥10% and ≥15% | Between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM group from Month 8 to Month 14 and between group differences for the Continue CGM and the Continue SMBG groups from baseline to Month 14 of proportion increasing
  Month 8 to Month 14 & Baseline to Month 14
Phase 2: Percent adding or removing diabetes medications | Month 8 to Month 14 & Baseline to Month 14
  Between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM group from Month 8 to Month 14 and between group differences for the Continue CGM and the Continue SMBG groups from baseline to Month 14 of percent adding or removing diabetes medications (starting or stopping medication)
Phase 2: Change in CGM glucose variability | Month 8 to Month 14 & Baseline to Month 14
  Between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM group from Month 8 to Month 14 and between group differences for the Continue CGM and the Continue SMBG groups from baseline to Month 14 of change in CGM glucose variability measured by the coefficient of variation
Phase 2: Change in CGM time-hypoglycemic | Month 8 to Month 14 & Baseline to Month 14
  Between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM group from Month 8 to Month 14 and between group differences for the Continue CGM and the Continue SMBG groups from baseline to Month 14 of change in CGM time-hypoglycemic, defined as <70mg/dL

OTHER OUTCOMES:
Phase 1 and Phase 2: Percent with glycated hemoglobin <7.0% | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2:Percent with glycated hemoglobin <7.5% | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Percent decreasing glycated hemoglobin by ≥1.0% (absolute) | Baseline to Month 8, Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  For Phase 1, the endpoints will be evaluated for between group differences in the CGM and SMBG groups from baseline to Month 8. For Phase 2, these endpoints will only be evaluated for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Percent decreasing glycated hemoglobin by ≥1.0% (absolute) OR reaching target glycated hemoglobin (<7.0%) | Baseline to Month 8, Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  For Phase 1, the endpoints will be evaluated for between group differences in the CGM and SMBG groups from baseline to Month 8. For Phase 2, these endpoints will only be evaluated for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Percent decreasing glycated hemoglobin by ≥10% (relative) | Baseline to Month 8, Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  For Phase 1, the endpoints will be evaluated for between group differences in the CGM and SMBG groups from baseline to Month 8. For Phase 2, these endpoints will only be evaluated for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Change in time <54 mg/dL | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Proportion of patients with time in target range ≥70% at Month 8 | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Change in the rate of CGM-measured hypoglycemic events | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  A CGM-measured hypoglycemic event is defined as at least 2 sensor values <54 mg/dL that are 15 or more minutes apart plus no intervening values >54 mg/dL; at least 2 sensor values >70 mg/dL that are 30 or more minutes apart with no intervening values ≤70 mg/dL, are required to define the end of an event, at which point the study patient becomes eligible for a new event.
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Change in time >180 mg/dL | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Change in time 300 mg/dL | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Area under curve 180 mg/dL | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Change in self-monitoring blood glucose frequency (self reported and download) | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Change in total daily insulin units per kg | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Change in basal units per kg | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Addition of at least one prandial insulin | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Addition of at least one GLP-1 analog or SGLT2 inhibitor | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Change in body weight | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Change in body mass index | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Change in blood pressure (systolic and diastolic blood pressure) | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Change in non HDL cholesterol | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: CGM use frequency (CGM group only) | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Questionnaires - Diabetes Distress Scale | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  Change in mean score and 4 subscales. Scored on a scale of 1 to 6. Higher scores mean a worse outcome.
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Questionnaires - Glucose Monitoring Satisfaction Survey | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  Change in mean score and 4 subscales.
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Questionnaires - Modified Hill-Bone Medication Adherence Scale | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  Change in total score. Scored on a scale of 8 to 32. Higher scores mean a worse outcome.
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Questionnaires - Clinician Communication Rating Scale | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  Change in mean score on 1 subscale. Scored on a scale of 1 to 4. Higher scores mean a better outcome.
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Questionnaires - Modified Toobert's Scale | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  Change in mean score. Scored on a scale of 0 to 7. Higher scores mean a better outcome.
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Questionnaires - Fear of Hypoglycemia Survey | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  Change in mean score. Scored on a scale of 0 to 4. Higher scores mean a worse outcome.
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Questionnaires - SF12 Health Survey | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  Change in Physical Health Composite score and Mental Health Composite score. Scored on a scale of 0 to 100. Higher scores mean a better outcome.
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Questionnaires - WHO-5 Well-Being Index | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  Change in total score.
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Questionnaires - CGM Satisfaction Survey | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  Given only to the CGM groups at follow-up so no comparison between groups. Scored on a scale from 0 to 100. Higher scores mean a better outcome.
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Questionnaires - Perceived Benefit Questionnaire | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  Given at follow-up only - Each item will be summarized individually; no total or mean score. There is no scale for this questionnaire.
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Questionnaires - Subjective Numeracy Scale | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  Given at study entry only so no comparison between groups. Scored on a scale of 1 to 6. Higher scores mean a better outcome.
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Safety Events - All adverse events | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Safety Events - Serious adverse events | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Safety Events - Severe hypoglycemia (defined as an event that required assistance from another person to administer carbohydrates or other resuscitative action) | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Safety Events - Diabetic ketoacidosis | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.
Phase 1 and Phase 2: Safety Events - Other adverse events | Baseline to Month 8, Month 8 to Month 14 & Baseline to Month 14
  The endpoints are the same for Phase 1 and Phase 2 and will only be listed once.
  Phase 1, between group differences in the CGM and SMBG groups from baseline to Month 8. Phase 2, between group differences for the Discontinue CGM Group (use SMBG only) and the Continue CGM Group from Month 8 to Month 14 as well as for the Continue CGM and the Continue SMBG groups from baseline to Month 14.

CONTACTS AND LOCATIONS:
Overall Officials: David Price, MD, Study Director — DexCom, Inc.
Locations (15):
- United States (15):
  - Keck School of Medicine @ USC, Los Angeles, California
  - Scripps Whittier Diabetes Institute, San Diego, California
  - Emory University, Atlanta, Georgia
  - Northwestern Memorial, Chicago, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - University of Michigan Internal Medicine, Ann Arbor, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - Park Nicollet International Diabetes Center, Minneapolis, Minnesota
  - Washington University Barnes Jewish Hospital, St Louis, Missouri
  - Las Vegas Endocrinology, Henderson, Nevada
  - University of North Carolina, Chapel Hill, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Lucas Research / Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - Vanderbilt Eskind Diabetes Clinic, Nashville, Tennessee
  - Amarillo Medical Specialists, LLP, Amarillo, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martens TW, Beck RW, Griffen C, Di J, Elkind-Hirsch K, Johnson ML, Castle JR, Beck SE, Bergenstal RM. Rapid improvements in glycemic management with use of continuous glucose monitoring in adults with type 2 diabetes treated with basal insulin: 3-month analysis of the MOBILE study. BMJ Open Diabetes Res Care. 2025 Nov 4;13(6):e005469. doi: 10.1136/bmjdrc-2025-005469. PMID 41192933
- [Derived] Davis G, Bailey R, Calhoun P, Price D, Beck RW. Magnitude of Glycemic Improvement in Patients with Type 2 Diabetes Treated with Basal Insulin: Subgroup Analyses from the MOBILE Study. Diabetes Technol Ther. 2022 May;24(5):324-331. doi: 10.1089/dia.2021.0489. Epub 2022 Apr 26. PMID 34962151
- [Derived] Bailey R, Calhoun P, Chao C, Walker TC. With or Without Residual C-Peptide, Patients with Type 2 Diabetes Realize Glycemic Benefits from Real-Time Continuous Glucose Monitoring. Diabetes Technol Ther. 2022 Apr;24(4):281-284. doi: 10.1089/dia.2021.0384. Epub 2022 Mar 21. PMID 34704817
- [Derived] Aleppo G, Beck RW, Bailey R, Ruedy KJ, Calhoun P, Peters AL, Pop-Busui R, Philis-Tsimikas A, Bao S, Umpierrez G, Davis G, Kruger D, Bhargava A, Young L, Buse JB, McGill JB, Martens T, Nguyen QT, Orozco I, Biggs W, Lucas KJ, Polonsky WH, Price D, Bergenstal RM; MOBILE Study Group; Type 2 Diabetes Basal Insulin Users: The Mobile Study (MOBILE) Study Group:. The Effect of Discontinuing Continuous Glucose Monitoring in Adults With Type 2 Diabetes Treated With Basal Insulin. Diabetes Care. 2021 Dec;44(12):2729-2737. doi: 10.2337/dc21-1304. Epub 2021 Sep 29. PMID 34588210
- [Derived] Martens T, Beck RW, Bailey R, Ruedy KJ, Calhoun P, Peters AL, Pop-Busui R, Philis-Tsimikas A, Bao S, Umpierrez G, Davis G, Kruger D, Bhargava A, Young L, McGill JB, Aleppo G, Nguyen QT, Orozco I, Biggs W, Lucas KJ, Polonsky WH, Buse JB, Price D, Bergenstal RM; MOBILE Study Group. Effect of Continuous Glucose Monitoring on Glycemic Control in Patients With Type 2 Diabetes Treated With Basal Insulin: A Randomized Clinical Trial. JAMA. 2021 Jun 8;325(22):2262-2272. doi: 10.1001/jama.2021.7444. PMID 34077499